CLINICAL TRIAL: NCT02866864
Title: Sensitization to Animal Allergens and Allergic Symptoms During Exposure to Animal Allergens in Korean Veterinary Researcher
Brief Title: Animal Allergy in Korean Veterinary Researcher
Status: Completed | Type: Observational
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Sang Min Lee, Assistant professor, Gachon University Gil Medical Center
Other Study IDs: GachonUGilMC
Record Dates: First submitted 2016-07-31; First posted 2016-08-15 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Rhinitis, Allergic; Asthma; Dermatitis, Atopic; Urticaria
Keywords: Allergen; Veterinary; Allergy; Animals
MeSH Terms: conditions — Rhinitis, Allergic; Asthma; Dermatitis, Atopic; Urticaria; Hypersensitivity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Subjects with animal allergy: Subjects who suffer from allergic symptom during contact with animal
  Interventions: Other: Animal allergy +
- Subjects without animal allergy: Subjects who do not suffer from allergic symptom during contact with animal
  Interventions: Other: Animal allergy -

INTERVENTIONS:
Other: Animal allergy + — Allergic symptom occurs when subject contact animal
  Groups: Subjects with animal allergy
Other: Animal allergy - — Allergic symptom does not occur when subject contact animal
  Groups: Subjects without animal allergy

SUMMARY:
The investigators will evaluate sensitization to animal allergens and allergic symptom during contacting animal allergens in Korean veterinary researchers who attend their annual conference.

The investigators will compare sensitization to animal allergen and other clinical and occupational factors between subjects who suffer from allergic symptom during contacting animal and those who do not.

DETAILED DESCRIPTION:
The investigators will visit annual conference of Korean veterinary researchers.

After informed consent, Korean veterinary researchers who attend their conference and agree to enrollment into this study will be asked to respond to questionnaires regarding their gender, age, underlying allergic diseases, family history of allergic diseases, occupation and it's duration, contact animal and contact duration. Subjects will also be requested to report allergic symptom, causal animal and situation of contact including veterinary service, animal experiment, pet ownership, and ingestion if subjects suffer from allergic symptom when subjects contact animal.

Then, subjects will also be asked to undergo skin prick test for animal allergens including chicken feather and ten mammal epithelia as well as cow's milk, and hen's egg, four fish flesh and seven animal meats.

subjects will be divided into two group, subjects who suffer from allergic symptom during contacting animal and those who do not. Between two groups, sensitization to animal allergens as well as other demographic and occupational factors including gender, age, underlying allergic diseases, family history of allergic diseases, occupation and it's duration, contact animal and contact duration will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Veterinary researchers attending their annual conference

Exclusion Criteria:

* Veterinary researchers who receive medication including antihistamine (H1 and H2 blocker), systemic glucocorticosteroid which can effect on the result of skin prick test
* Veterinary researchers who do not want to participate in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Korean Veterinary Researcher
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2016-08-26 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Skin reactivity to animal allergen in skin prick test | on the day of survey (day 1)
  Mean diameter of wheal for animal allergen in skin prick test

SECONDARY OUTCOMES:
Underlying allergic disease | on the day of survey (day 1)
  Underlying allergic disease including allergic rhinitis, asthma, atopic dermatitis, urticaria, food and drug allergy
Family history of allergic disease | on the day of survey (day 1)
  Family history of allergic disease including allergic rhinitis, asthma, atopic dermatitis, urticaria, food and drug allergy
Occupation | on the day of survey (day 1)
  Type of occupation including veterinary service and veterinary experiment
Duration of occupation | on the day of survey (day 1)
  Duration of occupation (year)
Contact animal | on the day of survey (day 1)
  Kinds of animals that subjects contact
Contact time | on the day of survey (day 1)
  Duration of animal contact (hour/day)
Causal animal | on the day of survey (day 1)
  Animal that provokes allergic symptom when subject contact it
Contact situation | on the day of survey (day 1)
  Situation including veterinary service, veterinary research, ingestion and pet ownership in which subject contact animal that provokes allergic symptom
Allergic symptom during contacting animal | on the day of survey (day 1)
  Allergic symptom including itchy eyes, nose and skin, rhinorrhea, sneezing, nasal congestion, postnasal drip, dyspnea, wheezing, cough, sputum, chest pain or discomfort, urticaria, rash, and angioedema when subject contact animal

CONTACTS AND LOCATIONS:
Overall Officials: Sang Min Lee, MD, PhD, Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant will be informed of results of questionnaires and skin prick test immediately after they complete questionnaires and skin prick test

REFERENCES:
- [Background] Blair A, Hayes HM Jr. Cancer and other causes of death among U.S. veterinarians, 1966-1977. Int J Cancer. 1980 Feb 15;25(2):181-5. doi: 10.1002/ijc.2910250203. PMID 7390647
- [Background] Elbers AR, Blaauw PJ, de Vries M, van Gulick PJ, Smithuis OL, Gerrits RP, Tielen MJ. Veterinary practice and occupational health. An epidemiological study of several professional groups of Dutch veterinarians. I. General physical examination and prevalence of allergy, lung function disorders, and bronchial hyperreactivity. Vet Q. 1996 Dec;18(4):127-31. doi: 10.1080/01652176.1996.9694711. PMID 8972059
- [Background] Samadi S, Spithoven J, Jamshidifard AR, Berends BR, Lipman L, Heederik DJ, Wouters IM. Allergy among veterinary medicine students in The Netherlands. Occup Environ Med. 2012 Jan;69(1):48-55. doi: 10.1136/oem.2010.064089. Epub 2011 May 31. PMID 21632519
- [Background] Park YB, Mo EK, Lee JY, Kim JH, Kim CH, Hyun IG, Choi JH. Association between pet ownership and the sensitization to pet allergens in adults with various allergic diseases. Allergy Asthma Immunol Res. 2013 Sep;5(5):295-300. doi: 10.4168/aair.2013.5.5.295. Epub 2013 Jun 25. PMID 24003386
- [Result] Moghtaderi M, Farjadian S, Abbaszadeh Hasiri M. Animal allergen sensitization in veterinarians and laboratory animal workers. Occup Med (Lond). 2014 Oct;64(7):516-20. doi: 10.1093/occmed/kqu097. Epub 2014 Aug 7. PMID 25104279
- [Result] Lutsky I, Baum GL, Teichtahl H, Mazar A, Aizer F, Bar-Sela S. Occupational respiratory disease in veterinarians. Ann Allergy. 1985 Aug;55(2):153-6. PMID 4025958
- [Result] Susitaival P, Kirk JH, Schenker MB. Atopic symptoms among California veterinarians. Am J Ind Med. 2003 Aug;44(2):166-71. doi: 10.1002/ajim.10253. PMID 12874849
- [Result] Krakowiak A, Wiszniewska M, Krawczyk P, Szulc B, Wittczak T, Walusiak J, Palczynski C. Risk factors associated with airway allergic diseases from exposure to laboratory animal allergens among veterinarians. Int Arch Occup Environ Health. 2007 May;80(6):465-75. doi: 10.1007/s00420-006-0153-0. Epub 2006 Oct 5. PMID 17021840
- [Result] Will LA, Nassif EG, Engen RL, Patterson RA, Zimmerman D. Allergy and pulmonary impairment in Iowa veterinarians. N Engl Reg Allergy Proc. 1987 May-Jun;8(3):173-7. doi: 10.2500/108854187778984645. PMID 3477686
- [Result] Samadi S, Wouters IM, Heederik DJ. A review of bio-aerosol exposures and associated health effects in veterinary practice. Ann Agric Environ Med. 2013;20(2):206-21. PMID 23772565